CLINICAL TRIAL: NCT04936763
Title: A Multicentre, Open-Label, Interventional, Trial To Assess The Performance And Tolerance Of Janesse 20 In The Volume Restoration Of Labia Majora
Brief Title: To Assess The Performance And Tolerance Of Janesse 20 In The Volume Restoration Of Labia Majora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0619/MD
Record Dates: First submitted 2021-05-31; First posted 2021-06-23 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Dysmorphic Disorder (BDD); Congenital Labia Majora Hypotrophy; Post-menopausal Labia Majora Hypotrophy
Keywords: Labia Majora; Genital rejuvenation; Hyaluronic Acid; Filler
MeSH Terms: conditions — Brachydactyly, Type D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Janesse 20 (Experimental)
  Interventions: Device: Janesse 20 (Cross-linked Hyaluronic Acid)

INTERVENTIONS:
Device: Janesse 20 (Cross-linked Hyaluronic Acid) — Janesse 20 will be administered at baseline (visit 2, day 0) and, if the Investigator will evaluate necessary, also at day 30 (visit 3). The Investigational device will be injected with retrograde technique (moving backward) with homogeneous amount on the length of each side of Labia Majora. The Janesse 20 dosage administered will be 1 ml in left labia and 1 ml in right labia for each session.

SUMMARY:
The use of hyaluronic acid (HA)-based fillers administered by injection to obtain Labia Majora augmentation is performed by many surgeons and gynaecologists in Europe, US and other countries, but few studies have investigated the effectiveness of this procedure. In this open not comparative study, 36 female subjects above or equal to 18 years old at inclusion, seeking genital rejuvenation, who have congenital or post-menopausal hypotrophy of the vulvar Labia Majora (or a diagnosis of Body Dysmorphic Disorder), who have given her informed consent and meet all the eligibility criteria, will be enrolled. Subjects will come to a total of 4 visits over a period of 2 months.

The primary objective of the study is to evaluate the performance of the dermal filler by the Global Aesthetic Improvement Scale (GAIS) at day 60 and the safety during all the study. The secondary objectives are the evaluation of volume restoration of Labia Majora (measured by caliper and Ultrasound) and the subjective evaluation (by Genital Appearance Satisfaction Scale) at different visits.

ELIGIBILITY:
Inclusion Criteria:

* Women with age ≥ 18.
* Women seeking genital rejuvenation with Genital Appearance Satisfaction Scale (GAS) >20 and Cosmetic Procedure Screening Scale modified for Labia (COPS-L)>40 .
* Patients with diagnosis of Body Dysmorphic Disorder (BDD) following DSM-IV criteria or congenital or post-menopausal Labia Majora hypotrophy
* • The Labia Majora (left and right) width and/or length must be between the 5th and 95th percentiles as reported in the Annex 4 of the protocol (modified table from Kreklau A e t al 2018). The measurement must be performed by the Investigators using the Sliding Zuricher Caliper mm130.
* Women willing to provide signed informed consent to clinical investigation participation.

Exclusion Criteria:

* Use of aspirin and antiplatelet agents a week prior to treatment.
* Pregnant or lactating women.
* Women with history of allergy or hypersensitivity to the HA or to other ingredients of the dermal filler.
* Women with history of allergy or hypersensitivity to Lidocaine, Mepivacaine or Prilocaine or local anaesthetics.
* Women with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma etc.
* Women presenting bleeding disorders in the past or present.
* Women taking or having indications for anticoagulant therapy.
* Use of concomitant treatments or procedures aimed to improve genital skin rejuvenation over the last six months before the clinical investigation enrolment, such as chemical peeling, dermabrasion, laser resurfacing.
* Women suffering from infectious diseases including herpes simplex virus infection, active hepatitis, Human Papilloma Virus (HPV) or Human Immunodeficiency Virus (HIV).
* Women suffering from local dermatitis (vulvar scaly papilloma, mycosis, bacterial infection near the injection area).
* Women at risk in term of precautions, warnings and contra-indications referred in the package insert of the clinical investigation device.
* Women with autoimmune diseases, streptococcus disease.
* Women with any active irritation or inflammation in the target areas of injection.
* Recent vulvae surgery in the treatment area or progressive recent or nearby cancers (i.e. cervical cancer).
* Tachycardia or other severe heart rhythm disorders
* Women with previous regional radiotherapy.
* Women who practice cycling or dedicate themselves to horse riding; women who practice bodybuilding or who perform professional sports.
* Women unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits.
* Performed dentist visit in the last week.
* Women participating in another clinical investigation or treated with another HA filler with the same indications at the same time or within the preceding 30 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women seeking genital rejuvenation with Genital Appearance Satisfaction Scale (GAS) >20
Enrollment: 36 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | 60 days
  Global Aesthetic Improvement Scale (GAIS) is will be evaluated by the investigator using standardized photos. The scale is using scores as 1= VERY MUCH IMPROVED, 2= MUCH IMPROVED, 3 = IMPROVED, 4 = NO CHANGE, 5= WORSE.
  The picture will be done at 60 days after the initiation of treatment with Janesse 20, will be compared with Baseline Visit (day 0) and one of the above-mentioned scores will be gibed used to indicate the changes after the treatment.
Overall safety | up to 60 days
  The overall safety will be evaluated by safety checklist for the patient (modified from Liu S, 2010) and the searching of Adverse Event (s), Adverse Device Event (s), Serious Adverse Event (s), Serious Adverse Device Event (s), Unanticipated Serious Adverse Device Event (s) and Device Deficiency at each visit.

SECONDARY OUTCOMES:
Dimensions of Labia Majora | 30 days, 60 days
  The measurement will be performed with the subject in lithotomy position at the different visits using a Sliding Zuricher Caliper mm130 for length and width; the ultrasound technique will be used to evaluate the depth.
Genital Appearance Satisfaction (GAS) | 30 days, 60 days
  Genital Appearance Satisfaction (GAS) self-assessment of the subject to assess the change comparing the final and baseline value. The scale contains 11 statements regarding attitudes towards genital appearance. Each item is scored on a Likert scale between 0 (="NEVER") and 3 =("ALWAYS"). Total scores range from 0 to 33. Higher scores represent greater dissatisfaction with the genitalia.
Global Aesthetic Improvement Scale (GAIS) | 30 days, 60 days
  Global Aesthetic Improvement Scale (GAIS) evaluated by blind Investigator, using scores 1= VERY MUCH IMPROVED, 2= MUCH IMPROVED, 3 = IMPROVED, 4 = NO CHANGE, 5= WORSE.

OTHER OUTCOMES:
Explorative outcome (Labia Majora volume) | 30 days, 60 days
  The validation of measurements of Labia Majora volume by a 3D software during the study period comparing these values with the dimensions obtained with ultrasound (for depth) and caliper (for lenght and width).
  Tridimensional surface imaging for estimating Labia Majora volume using Crisalix iPad App and the Crisalix 3D Surface Imager Camera will be evaluated by blind Investigator at different visits. The data will be collected and evaluated in 1 center only (Genova).

CONTACTS AND LOCATIONS:
Locations (2):
- Villa Serena, Genova, Italy
- SCM Dr Rosu, Timișoara, Romania

REFERENCES:
- [Background] Cosmetic Surgery National Data Bank Statistics. Aesthet Surg J. 2017 May 1;37(suppl_2):1-29. doi: 10.1093/asj/sjx076. No abstract available. PMID 28388734
- [Background] Bucknor A, Chen AD, Egeler S, Bletsis P, Johnson AR, Myette K, Lin SJ, Hamori CA. Labiaplasty: Indications and Predictors of Postoperative Sequelae in 451 Consecutive Cases. Aesthet Surg J. 2018 May 15;38(6):644-653. doi: 10.1093/asj/sjx241. PMID 29342228
- [Background] Ouar N, Guillier D, Moris V, Revol M, Francois C, Cristofari S. [Postoperative complications of labia minora reduction. Comparative study between wedge and edge resection]. Ann Chir Plast Esthet. 2017 Jun;62(3):219-223. doi: 10.1016/j.anplas.2017.02.005. Epub 2017 Mar 9. French. PMID 28285885
- [Background] Vanaman M, Bolton J, Placik O, Fabi SG. Emerging Trends in Nonsurgical Female Genital Rejuvenation. Dermatol Surg. 2016 Sep;42(9):1019-29. doi: 10.1097/DSS.0000000000000697. PMID 27153040
- [Background] Hunter JG. Labia Minora, Labia Majora, and Clitoral Hood Alteration: Experience-Based Recommendations. Aesthet Surg J. 2016 Jan;36(1):71-9. doi: 10.1093/asj/sjv092. Epub 2015 Oct 24. PMID 26499942
- [Background] Sharp G, Mattiske J, Vale KI. Motivations, Expectations, and Experiences of Labiaplasty: A Qualitative Study. Aesthet Surg J. 2016 Sep;36(8):920-8. doi: 10.1093/asj/sjw014. Epub 2016 Feb 23. PMID 26912581
- [Background] Sorice SC, Li AY, Canales FL, Furnas HJ. Why Women Request Labiaplasty. Plast Reconstr Surg. 2017 Apr;139(4):856-863. doi: 10.1097/PRS.0000000000003181. PMID 28350660
- [Background] Sharp G, Tiggemann M, Mattiske J. Factors That Influence the Decision to Undergo Labiaplasty: Media, Relationships, and Psychological Well-Being. Aesthet Surg J. 2016 Apr;36(4):469-78. doi: 10.1093/asj/sjv270. Epub 2016 Feb 18. PMID 26893523
- [Background] Goodman MP, Placik OJ, Benson RH 3rd, Miklos JR, Moore RD, Jason RA, Matlock DL, Simopoulos AF, Stern BH, Stanton RA, Kolb SE, Gonzalez F. A large multicenter outcome study of female genital plastic surgery. J Sex Med. 2010 Apr;7(4 Pt 1):1565-77. doi: 10.1111/j.1743-6109.2009.01573.x. Epub 2009 Nov 12. PMID 19912495
- [Background] Veale D, Eshkevari E, Ellison N, Costa A, Robinson D, Kavouni A, Cardozo L. A comparison of risk factors for women seeking labiaplasty compared to those not seeking labiaplasty. Body Image. 2014 Jan;11(1):57-62. doi: 10.1016/j.bodyim.2013.10.003. Epub 2013 Nov 14. PMID 24239491
- [Background] Jackson TD, Grilo CM, Masheb RM. Teasing history, onset of obesity, current eating disorder psychopathology, body dissatisfaction, and psychological functioning in binge eating disorder. Obes Res. 2000 Sep;8(6):451-8. doi: 10.1038/oby.2000.56. PMID 11011912
- [Background] de Jong PJ, van Overveld M, Schultz WW, Peters ML, Buwalda FM. Disgust and contamination sensitivity in vaginismus and dyspareunia. Arch Sex Behav. 2009 Apr;38(2):244-52. doi: 10.1007/s10508-007-9240-x. Epub 2007 Oct 2. PMID 17909958
- [Background] Hamori CA. Discussion: Why Women Request Labiaplasty. Plast Reconstr Surg. 2017 Apr;139(4):864. doi: 10.1097/PRS.0000000000003183. No abstract available. PMID 28350661
- [Background] Berreni N. Augmentation of the Labia Majora With Fillers. In: Hamori CA, Banwel PE, Alinsod R, editors. Female Cosmetic Genital Surgery: concepts, classification, and techniques. New York: Thieme Medical Publishers, Inc; 2017. p 125-142.
- [Background] Jabbour S, Kechichian E, Hersant B, Levan P, El Hachem L, Noel W, Nasr M. Labia Majora Augmentation: A Systematic Review of the Literature. Aesthet Surg J. 2017 Oct 16;37(10):1157-1164. doi: 10.1093/asj/sjx056. PMID 28449124
- [Background] Fasola E, Gazzola R. Labia Majora Augmentation with Hyaluronic Acid Filler: Technique and Results. Aesthet Surg J. 2016 Nov;36(10):1155-1163. doi: 10.1093/asj/sjw083. Epub 2016 May 30. PMID 27241363
- [Background] Hexsel D, Dal'Forno T, Caspary P, Hexsel CL. Soft-Tissue Augmentation With Hyaluronic Acid Filler for Labia Majora and Mons Pubis. Dermatol Surg. 2016 Jul;42(7):911-4. doi: 10.1097/DSS.0000000000000733. No abstract available. PMID 27227470
- [Background] Zerbinati N, Haddad RG, Bader A, Rauso R, D'Este E, Cipolla G, Calligaro A, Gonzalez P, Salvatore S, Serafin D. A new hyaluronic acid polymer in the augmentation and restoration of labia majora. J Biol Regul Homeost Agents. 2017 APR-JUN;31(2 Suppl. 2):153-161. PMID 28702976
- [Background] Bramwell, R, Morland, C. Genital appearance satisfaction in women: The development of a questionnaire and exploration of correlates. Journal of Reproductive and Infant Psychology. 2009; 27, 15-27.
- [Background] Veale D, Eshkevari E, Ellison N, Cardozo L, Robinson D, Kavouni A. Validation of genital appearance satisfaction scale and the cosmetic procedure screening scale for women seeking labiaplasty. J Psychosom Obstet Gynaecol. 2013 Mar;34(1):46-52. doi: 10.3109/0167482X.2012.756865. PMID 23394414
- [Background] Kreklau A, Vaz I, Oehme F, Strub F, Brechbuhl R, Christmann C, Gunthert A. Measurements of a 'normal vulva' in women aged 15-84: a cross-sectional prospective single-centre study. BJOG. 2018 Dec;125(13):1656-1661. doi: 10.1111/1471-0528.15387. Epub 2018 Aug 1. PMID 29940085
- [Background] Lindqvist C, Tveten S, Bondevik BE, Fagrell D. A randomized, evaluator-blind, multicenter comparison of the efficacy and tolerability of Perlane versus Zyplast in the correction of nasolabial folds. Plast Reconstr Surg. 2005 Jan;115(1):282-9. PMID 15622265
- [Background] Fasola E, Bosoni D. Dynamic Quadripolar Radiofrequency: Pilot Study of a New High-Tech Strategy for Prevention and Treatment of Vulvar Atrophy. Aesthet Surg J. 2019 Apr 8;39(5):544-552. doi: 10.1093/asj/sjy180. PMID 30052757
- [Background] Joumblat NR, Chim J, Aguirre Sanchez PG, Bedolla E, Salgado CJ. Guidelines for the Standardization of Genital Photography. Aesthet Surg J. 2018 Sep 14;38(10):1124-1130. doi: 10.1093/asj/sjy017. PMID 29420725
- [Background] EHRENPREIS S, KELLOCK MG. The interaction of quarternary ammonium compounds with hyaluronic acid. Biochim Biophys Acta. 1960 Dec 18;45:525-8. doi: 10.1016/0006-3002(60)91489-x. No abstract available. PMID 13725990
- [Background] Georgiev GA, Yokoi N, Ivanova S, Dimitrov T, Andreev K, Krastevd R, Lalcheva Z. Surface chemistry study of the interactions of hyaluronic acid and benzalkonium chloride with meibomian and corneal cell lipids. Soft Matter, 2013,9, 10841-10856.
- [Background] Liu S, Ercolano E, Siefert ML, McCorkle R. Patterns of symptoms in women after gynecologic surgery. Oncol Nurs Forum. 2010 Mar;37(2):E133-40. doi: 10.1188/10.ONF.E133-E140. PMID 20189912
- [Background] Migda MS, Migda M, Slapa R, Mlosek RK, Migda B. The use of high-frequency ultrasonography in the assessment of selected female reproductive structures: the vulva, vagina and cervix. J Ultrason. 2019 Dec;19(79):261-268. doi: 10.15557/JoU.2019.0039. Epub 2019 Dec 31. PMID 32021707